CLINICAL TRIAL: NCT04476563
Title: Checkpoint Inhibitor-induced Liver Injury Study (ChILI)
Brief Title: Checkpoint Inhibitor-induced Liver Injury
Acronym: ChILI
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20034
Record Dates: First submitted 2020-07-02; First posted 2020-07-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Immune-Mediated Hepatitis
Keywords: Immune checkpoints inhibitors; Immune-related adverse events; Hepatotoxicity; Liver injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Collection and storage of biological samples (blood, urine, stool) from patients with ChILI at three-time points (the day of liver injury, 1 week, and 1 month after). The investigators will perform a liver biopsy when it is clinically indicated.
  * Collection and storage of biological samples (blood, urine, and stool) from control patients at two-time points (before starting CPIs and 6 to14 weeks after commencing treatment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ChILI: Patients who are already on CPI therapy and have developed liver injury
  Interventions: Diagnostic Test: Obtaining biological samples
- Control: Patients with cancer who are starting on checkpoint inhibitors
  Interventions: Diagnostic Test: Obtaining biological samples

INTERVENTIONS:
Diagnostic Test: Obtaining biological samples — Biological samples (blood, urine, stool). Liver tissue will be obtained from ChILI group when clinically indicated

SUMMARY:
In this multi-center prospective observational study, the investigators plan to identify the incidence and risk factors for checkpoint inhibitor-induced liver injury and characterize biochemical, genetic, immunological, and histological features associated with it.

DETAILED DESCRIPTION:
Checkpoint inhibitor-induced liver injury (ChILI) is a new incompletely understood category of hepatotoxicity which is distinct from other types of drug-induced liver injury (DILI) such as direct or idiosyncratic DILI. The data regarding the incidence and risk factors is lacking. Therefore, 'in-depth phenotyping' together with data from the control group exposed to checkpoint inhibitors (CPI) is necessary to develop refined algorithms incorporating CPI-related factors, host genetic and environmental risk factors that would enable pre-empting ChILI.

The aim of the study is to enroll two deeply phenotyped cohorts (patients who developed ChILI and patients who are starting checkpoint inhibitors) and obtain biological samples at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

Both patient groups and control group:

• Able to give written informed consent OR Potential participants who have developed encephalopathy related to ChILI as a response to checkpoint inhibitor therapy, who lack the capacity to give written informed consent and have a consultee (personal or nominated) - for ChILI patient group only

ChILI group:

Patients who developed checkpoint inhibitor-induced liver injury and meet the following criteria:

1. Meets one of the following analytical thresholds at enrolment (visit 1)

   * Alanine transaminase (ALT) exceeding 5 times the upper limit of normal (ULN) OR
   * ALT exceeding 3 times ULN plus bilirubin exceeding 2 times ULN OR
   * Alkaline phosphatase (ALP) exceeding 2 times ULN with accompanying elevations of gamma-glutamyl transferase in the absence of known bone metastases driving the rise in ALP level
2. Absence of other known causes of liver injury after detailed investigations

Patients who developed ChILI but did not meet the above criteria at enrolment or who were found to have a different cause for their liver injury after further investigations will be excluded from the analysis

Control group:

Consecutive patients with cancer who have a clinical indication to start checkpoint inhibitors. A small proportion of patients will develop ChILI following their checkpoint inhibitor treatment and will be classified as cases.

Exclusion Criteria:

* Patients who are treated with cytotoxic chemotherapy concurrently with checkpoint inhibitors.
* On the judgment of chief investigator that the person has certain alternative explanations to the acute event (rather than ChILI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ChILI group:
  Adults with cancer receiving checkpoint inhibitors (CTLA-4, PD-1 or PD L1 inhibitor) as monotherapy or combination (without chemotherapy) and developed acute liver injury secondary to checkpoint inhibitor.
  Control Group:
  Patients with malignant melanoma, renal cell carcinoma, non-small cell lung cancer or any other cancer, receiving single or combination therapy using checkpoint inhibitors (CPIs).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of checkpoint inhibitor-induced liver injury (ChILI) and other immune-mediated adverse reactions | 3 years
Identify novel biomarkers associated with the diagnosis of ChILI | 3 years
  The investigators plan assessment of proposed circulating biomarkers including cytokines, microRNAs (miR-122, miR-4270 and miR-4463), total cytokeratin 18 (K18), macrophage colony-stimulating factor receptor (MCSFR), and any others identified in subsequent publications and measure their diagnostic and prognostic accuracy using the area under the receiver operating curve (AUROC).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

REFERENCES:
- [Derived] Ji C, Kumpf S, Qian J, Federspiel JD, Sheehan M, Capunitan D, Atallah E, Astbury S, Arat S, Oziolor E, Ocana MF, Ramaiah SK, Grove J, Aithal GP, Lanz TA. Transcriptomic and proteomic characterization of cell and protein biomarkers of checkpoint inhibitor-induced liver injury. Cancer Immunol Immunother. 2025 May 3;74(6):190. doi: 10.1007/s00262-025-04033-z. PMID 40317333